CLINICAL TRIAL: NCT03730493
Title: A Study to Evaluate the Effectiveness of a Pictorial Flashcard Regarding Self-Care of Peripheral Intravenous Cannula (PIVC) on Its Indwelling Time and Related Complications Among Inpatients at ILBS, New Delhi
Brief Title: Effectiveness of a Pictorial Flashcard Regarding Self-care of Peripheral Intravenous Cannula (PIVC) on Its Indwelling Time and Related Complications Among Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Rahul Ranjan, Principal Investigator, Institute of Liver and Biliary Sciences, India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-01
Record Dates: First submitted 2018-10-13; First posted 2018-11-05 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Inpatient Facililty Diagnoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pictorial flashcard (Experimental): In the experimental group researcher explained self-care of PIVC using pictorial flashcard on one to one basis. Patients were explained Do's and Don'ts, they have to keep in mind during self-care. Doubts of the patients were also addressed simultaneously. After this a copy of pictorial flashcard was given to the subjects to be used in future (during PIVC in-situ). Time was noted and kept for observation till 72 hours or removal in between.
  Interventions: Behavioral: Teaching subjects regarding self-care of PIVC with Pictorial Flashcard.
- Comparison Group (No Intervention): In control group, standard care was given as per the hospital protocol.Time was noted and kept for observation till 72 hours or removal in between.

INTERVENTIONS:
Behavioral: Teaching subjects regarding self-care of PIVC with Pictorial Flashcard. — In the experimental group researcher explained self-care of PIVC using pictorial flashcard on one to one basis. Patients were explained Do's and Don'ts, they have to keep in mind during self-care or management. Doubts of the patients were also addressed simultaneously. After this a copy of pictorial flashcard was given to the subjects to be used in future (during PIVC in-situ). In control group, standard care was given as per the hospital protocol. After 24 hours/one day, PIVC was observed for presence of any complications such as Phlebitis, Infiltration, Pain, Blockage and Dislodgement using V.I.P. Score, Infusion nurses society infiltration scale, Universal pain assessment tool and PIVC Documentation Tool and need for PIVC removal was also assessed. After 72 hours PIVC removed (whatever applicable) site of PIVC was reassessed, reason for removal was recorded and indwelling time was noted.
  Arms: Pictorial flashcard

SUMMARY:
The study title is "A Study to evaluate the Effectiveness of a Pictorial Flashcard regarding Self-Care of Peripheral Intravenous Cannula (PIVC) on its indwelling time and related complications among inpatients at ILBS, New Delhi." and it aim to evaluate the Effectiveness of a Pictorial Flashcard regarding Self-Care of PIVC on its indwelling time and related complications among inpatients.

DETAILED DESCRIPTION:
Objectives of the Study

1. To evaluate the Effectiveness of a Pictorial Flashcard regarding Self-Care of PIVC on its indwelling time and related complications among inpatients.
2. To find out the association between indwelling time of PIVC with selected demographic and clinical variables.
3. To find out the association between PIVC related complications with selected demographic and clinical variables.

Setting of the Study General wards of ILBS, New Delhi

Population Inpatients with PIVC

Sampling Technique Convenient sampling technique.

Data collection Data will be collected from the study subjects as well as from medical records. Subjects were taken from General wards of Institute of Liver and Biliary Sciences, New Delhi.

Methodology Research Approach: Quantitative research approach. Research Design: Quasi Experimental Research design (Post-test only comparison group Design) Sample size: 80 (40 in each group), finalize after power analysis

Data Analysis Method Descriptive statistics: Mean, frequency, percentage distribution and Standard Deviation Inferential Statistics: Chi Square, t- test ANOVA, RM-ANOVA and Man-Whitney U test.

ELIGIBILITY:
Inclusion Criteria

Patients who:

* were conscious & oriented.
* could understand Hindi or English.
* were between the age group of 18 to 60 years.
* were admitted in general wards and scheduled for PIVC insertion
* received IV infusion and/or medication for at least 3 days (72 hours)

Exclusion Criteria

Patients who:

* were on physical restraints
* were on sedative drugs.
* in whom PIVC was removed for the sole purpose of discharge before 72 hours.
* had short admission period, i.e less than 72 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Pictorial Flashcard on Indwelling time of Peripheral Intravenous Cannula (PIVC) among inpatients. | 72 hours
  Effectiveness refers to the significant increase in indwelling time of PIVC and reduction in PIVC related complication after using pictorial flash card on self-care of PIVC which calculated in hours i.e. 72 hours.
  Indwelling time refers to the time duration i.e. 72 hours between insertion and removal of PIVC.
Adverse events (complications related to PIVC) in both groups. | 72 hours
  Adverse events or complications related to PIVC refers to complications, such as Phlebitis, Infiltration, Pain,Blockage and Dislodgement which occurs on PIVC site during the indwelling time of PIVC i.e. within or till 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No